CLINICAL TRIAL: NCT02029261
Title: Project 4: Molecular Mechanisms in Burn-induced Insulin Resistance in Humans
Brief Title: Observational Study of Insulin Resistance and Muscle Wasting After Burn Injury
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ronald G. Tompkins, Chief, Burns Division, Massachusetts General Hospital
Other Study IDs: P50GM021700P4_1; 2P50GM021700-32A1 (NIH)
Record Dates: First submitted 2013-12-17; First posted 2014-01-07 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Burn
Keywords: Burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, plasma, isolated leukocytes, skeletal muscle, fat, skin
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine important and significant problems, that of insulin resistance and muscle wasting after burn injury.

DETAILED DESCRIPTION:
Burn injury induces insulin resistance and our investigators have previous shown the importance of insulin receptor substrate 1 (IRS-1)-mediated pathways. This project will establish the inhibitory effects of burn injury on IRS-1 mediated signaling in human skeletal muscle of burn patients.

ELIGIBILITY:
Inclusion Criteria:

* Burn injury >=10% total body surface area involvement from any etiology that will require surgical treatment
* Age 18 years or older
* Admitted to the Massachusetts General Hospital within 30 days of burn injury
* Patient or guardian who is capable of giving full informed consent

Exclusion Criteria:

* Decision not to treat due to severity of injury
* Presence of anoxic brain injury that is not expected to result in complete recovery
* Existence of co-morbid conditions of malignancy currently under treatment, medical condition requiring glucocorticoid treatment, insulin dependent diabetes mellitus, morbid obesity defined as body mass index >= 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Massachusetts General Hospital (MGH) burn patients from the emergency department, intensive care unit, burn unit, or other MGH inpatient unit
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Determination of gene expression profile and protein expression | Time of burn injury up to 24 months postinjury
  Determination of individual profiles and comparison with profiles from existing patients and healthy controls

SECONDARY OUTCOMES:
Hospital discharge status | From hospital admission to discharge
  Alive or dead
Presence of clinical complications | From hospital admission to discharge
  Analysis of incidence of clinical complications related to organ function/dysfunction
Intensive care unit (ICU) days | From hospital admission to discharge
  Total number of ICU days
Nutritional status at discharge | At hospital discharge
  Analysis of change in total body weight, lean body mass, indirect calorimetry, and nitrogen balance
Correlation between protein data and in vivo physiologic measurement data | Hospitalization
  Gene and and protein expression data will be correlated with the physiological and and in vivo physiologic measurements (lab values) and nutritional status data.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Tompkins, MD, ScD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data provided to the journal as required for publication